CLINICAL TRIAL: NCT02863887
Title: The Lifestyle Changes Through Exercise and Nutrition (LEAN) Project
Brief Title: Lifestyle Changes Through Exercise and Nutrition
Acronym: LEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2016-018
Record Dates: First submitted 2016-07-07; First posted 2016-08-11 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Diabetes
Keywords: Weight Loss; African American; Community Based; Mobile technology; Translational science
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight loss intervention (Experimental): Churches randomized to the intervention condition will receive the community health coach delivered church based intervention for 6 months followed by 6 months of weight maintenance.
  Interventions: Behavioral: Weight loss intervention
- Delayed Treatment Control Group (Experimental): Churches in the delayed treatment control condition will receive information on various health topics relevant to African Americans, such as strokes, lupus, sickle cell, etc. via text message during the first six months. Participants in this group will not receive any behavioral strategies designed to alter weight, physical activity, or diet during this time. They will receive the community health coach delivered church based weight loss intervention after 6 months.
  Interventions: Behavioral: Weight loss intervention

INTERVENTIONS:
Behavioral: Weight loss intervention — The intervention will involve utilizing trained community health coaches to deliver the weight loss intervention. There will be 10 group based sessions conducted at each church over 6 months. Session frequency will be 4 weekly sessions (4) for the first month, bimonthly sessions for 2 months (4) and monthly sessions for 2 months (2). The study is based upon weight loss strategies that have been utilized in the Diabetes Prevention Program. The group sessions will be augmented by utilizing text messages. The text messages will be delivered weekly and three types of messages will be delivered: 1) lesson content, 2) motivational, 3) behavioral prompts.

SUMMARY:
The goal of The LEAN project intervention is to promote weight loss, healthy dietary habits, increased physical activity, improved blood glucose and cholesterol, and weight related quality of life in obese African American adults through a sustainable, technology enhanced, church-based program.

DETAILED DESCRIPTION:
The LEAN Project is a community-based weight loss program that is delivered through churches serving lower-income, obese, African American adults. The intervention will involve training community health coaches to deliver the intervention. These community health coaches will be individuals who are members of the church and who are willing to be trained on how to deliver behaviorally-based, empirically proven, lifestyle change interventions. These community health coaches will be trained by the staff at Pennington Biomedical, who have experience training and delivering these types of interventions. The community health coaches will deliver the intervention through their respective church after being trained. Weekly text messages will be sent to participants in order to supplement the intervention sessions and provide support. The primary aim is to determine if the trained community health coach church-based intervention will result in significant weight loss. Secondary aims will assess blood glucose, cholesterol, physical activity, food intake, and weight related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* a member of a participating church
* age 18-75 years old
* BMI > 30
* own a mobile phone with text message capabilities
* at risk for diabetes (diagnosed nuclear family member or gestational diabetes) or diagnosed with type 2 diabetes
* willing to provide written informed consent
* willing to change diet, physical activity and weight
* able to participate in face-face counselling sessions as scheduled
* low to moderate cardiovascular disease risk

Exclusion Criteria:

* currently participating in a weight loss program
* currently using weight loss medication or have lost weight (>10 lbs in last year)
* planning to move from the area within the next year
* given birth within the past year, are currently pregnant or plan to become pregnant within the next year
* planning to have bariatric surgery within 2 years
* history of major depression, suicidal behavior or eating disorder
* hospitalization for a mental disorder or substance abuse in the last year
* have cancer or had cancer within the past 5 years.
* serious heart problems such as arrhythmias, cardiomyopathy, congestive heart failure
* stroke or heart attack in the last six months
* high blood pressure [systolic ≥160, or diastolic ≥100]
* chronic inflammatory conditions, including but not limited to severe arthritis, lupus, or inflammatory bowel disease
* diseases that are life threatening or that can interfere with or be aggravated by exercise or weight loss
* unwilling or unable to provide informed consent
* physician's or principal investigator's decision to exclude

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09-23 (Actual); Study Completion 2017-09-23 (Actual)

PRIMARY OUTCOMES:
Percent weight loss | Month 6 and Year 1
  Percent weight loss will be calculated at 6 and 12 months.

SECONDARY OUTCOMES:
Change in Body Fat Percentage | Screening, Month 6 and Year 1
  The participant's body fat percentage is measured using the portable Tanita Body Composition Analyzer (SC-240).
Change in Blood Glucose | Screening, Month 6 and Year 1
  The Alere Cholestech LDX® Analyzer is engineered to provide accurate, actionable, and readily accessible glucose testing results. The Cholestech uses fingerstick sampling and small sample size (40μL) that makes results less time consuming and easy to obtain.
Change in Blood Pressure | Screening, Month 6 and Year 1
  Blood pressure will be measured using an automatic blood pressure cuff (Omeron, Model BP710 or similar). Participants will rest for approximately 5 minutes prior to blood pressure measurement to ensure accurate at rest reading.
Change in Food Intake | Screening, Month 6 and Year 1
  The National Cancer Institute (NCI) fat screener estimates the percentage of energy from fat by asking patients to report the frequency of consuming specific foods over the past 12 months. A standard 7-item fruit and vegetable screener developed by the NCI and National 5 a Day Program grantees asks how often fruit and vegetables were consumed in the past month.
Change in Physical activity | Screening, Month 6 and Year 1
  The International Physical Activity Questionnaire (IPAQ) questionnaire is a self-report measure of physical activity. The metabolic equivalent task (MET) minutes in each domain of leisure time activity, that is, sedentary, light, moderate, and vigorous intensity, will be calculated. The IPAQ has been shown to be a reliable and valid measure of physical activity and has been sensitive to changes in physical activity resulting from intervention programs.
Change in Quality of Life | Screening, Month 6 and Year 1
  . Each participant's quality of life will be assessed using the Impact of Weight on Quality of Life Survey.
Satisfaction Questionnaire | Month 6 and Year 1
  Each participant's satisfaction with the different elements of the study, including the community health coaches, the intervention, and the text messages, will be measured using a questionnaire developed by the investigators.
Change in Blood Cholesterol | Screening, Month 6 and Year 1
  The Alere Cholestech LDX® Analyzer is engineered to provide accurate, actionable, and readily accessible cholesterol testing results. The Cholestech uses fingerstick sampling and small sample size (40μL) that makes results less time consuming and easy to obtain.
Change in Pulse | Screening, Month 6 and Year 1
  Pulse will be measured using an automatic blood pressure cuff (Omeron, Model BP710 or similar). Participants will rest for approximately 5 minutes prior to pulse measurement to ensure accurate at rest reading.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Newton, Jr., PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen T, Irwin ML, Dewan AT, Cartmel B, Harrigan M, Ferrucci LM, Sanft T, Li F, Lu L, Salinas YD. Examining the effect of obesity-associated gene variants on breast cancer survivors in a randomized weight loss intervention. Breast Cancer Res Treat. 2021 Jun;187(2):487-497. doi: 10.1007/s10549-021-06151-5. Epub 2021 Mar 6. PMID 33677781
- [Derived] Newton RL Jr, Carter LA, Johnson W, Zhang D, Larrivee S, Kennedy BM, Harris M, Hsia DS. A Church-Based Weight Loss Intervention in African American Adults using Text Messages (LEAN Study): Cluster Randomized Controlled Trial. J Med Internet Res. 2018 Aug 24;20(8):e256. doi: 10.2196/jmir.9816. PMID 30143478